CLINICAL TRIAL: NCT02650492
Title: Exploratory Study on Immunostimulating Interstitial Laser Thermotherapy in Malignant Melanoma
Brief Title: Immunostimulating Interstitial Laser Thermotherapy in Malignant Melanoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped in agreement with investigator due to slow patient recruitment.
Sponsor: Clinical Laserthermia Systems AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-2015-004
Record Dates: First submitted 2015-11-27; First posted 2016-01-08 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Melanoma; Malignant Melanoma
Keywords: Hyperthermia, Induced; Laser Coagulation; Laser Therapy
MeSH Terms: conditions — Melanoma; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- imILT (Experimental): Immunostimulating Interstitial Laser Thermotherapy (imILT)
  Interventions: Device: Immunostimulating Interstitial Laser Thermotherapy

INTERVENTIONS:
Device: Immunostimulating Interstitial Laser Thermotherapy — Immunostimulating Interstitial Laser Thermotherpy (imILT) is a specific form of thermotherapy, which, in addition to destroying tumor tissue, has been optimized to cause a tumor specific immunologic response.

SUMMARY:
Thermotherapy is a technology aiming at destroying tissue, for example tumor tissue. Immunostimulating Interstitial Laser Thermotherpy (imILT) is a specific form of thermotherapy, which, in addition to destroying tumor tissue, has been optimized to cause a tumor specific immunologic response. In laboratory animals the imILT method has also been shown to induce a so called abscopal effect. This means that when one tumor is treated with imILT other, untreated, tumors also decrease in size. The immunologic response has previously been characterized in breast cancer patients after receiving imILT treatment , and presumed abscopal effects induced by imILT have also been described in a malignant melanoma patient.

The purpose of this trial is to investigate the functionality and safety of the imILT treatment method in patients diagnosed with malignant melanoma. The inflammatory process, following on the treatment, will also be described in order to provide a more in depth knowledge of the treatment for this indication. The purpose is also to evaluate efficiency when it comes to local tumor destruction as well as understanding of the subsequent immunological effects. Since immunologically based treatment of malignant melanoma is under intense review with so called "immune checkpoint inhibitors" this trial will also provide valuable information on how imILT, in the future, could be combined with these new and, for some patients, very effective treatment regimens.

The treatment method has successfully been used for treatment of patients with breast cancer and malignant melanoma . Treatment of breast cancer patients caused an increase of cytotoxic T lymphocytes in the treated tumor, as well as activated dendritic cells at the tumor border. Regulatory T lymphocytes decreased in the regional lymph nodes.

This trial is explorative, prospective, open and non-randomized. Five malignant melanoma patients stage III - IV will be treated in this trial, which is estimated to be carried out during a time period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* histologically confirmed malignant melanoma
* advanced melanoma disease (Stage III inoperable or Stage IV) that has progressed on standard first line treatment such as kinase inhibitor(s) and/or immunoregulatory monoclonal antibodies. Previously untreated patients with a dominant tumour lesion deemed suitable for local and highly tumour-destructive ablation may also be included
* time interval between previous systemic treatment and imILT of at least one month
* at least one lesion located in such a way (typically subcutaneously) that it can be treated without risk of skin necrosis or serious damage to other adjacent vital and healthy tissue
* verbal and written informed consent to participate
* adequate haematologic, renal and hepatic functions
* have an ECOG performance status ≤ 2 (Karnofsky ≥ 60%)

Exclusion Criteria:

* known HIV infection
* autoimmune disease which is judged to reduce an anti-tumour immune response
* systemic corticosteroid medication
* bleeding diathesis
* pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events) | 18 months
  Evaluation of adverse events.
Usability of the device as evaluated by treatment logs | 18 months
  Evaluation of the laser system by analysis of treatment logs of the device.
Usability of the device as evaluated by user questionnaire | 18 months
  Evaluation of the laser system by analysis of user questionnaire.

SECONDARY OUTCOMES:
Treatment effect (Measurement of tumor burden by irRC criteria) | 18 months
  Measurement of tumor burden by irRC criteria.
Inflammatory response in tumor and circulation measured by quantification of inflammatory cell populations | 18 months
  Quantification of cellular infiltrate and activation markers by immunohistochemistry and flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Hansson, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital Solna, Stockholm, Sweden